CLINICAL TRIAL: NCT02640040
Title: The Effect of Combined Surgery in Management of Congenital Pseudarthrosis of Tibia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Children's Hospital (Other Government)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan Women and Children's Medical Center (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Beijing Children's Hospital (Other); Dalian Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Kunming Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN02
Record Dates: First submitted 2015-08-31; First posted 2015-12-28 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Congenital Pseudarthrosis of Tibia
MeSH Terms: interventions — Fracture Fixation, Intramedullary; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- combined surgery (Experimental): combined surgery for enrolled patients with CPT(Congenital Pseudarthrosis of Tibia): sleeve resection of the pathological soft tissues, intramedullary rod fixation, packaged lilac bone autograft,and llizarov external fixation device installation.
  Interventions: Device: llizarov external fixation device; Device: intramedullary rod fixation; Procedure: surgery

INTERVENTIONS:
Device: llizarov external fixation device — llizarov external fixation device was applied to fix the tibia.
  Other Names: llizarov fixator
Device: intramedullary rod fixation — retrograde intramedullary rod was applied to stabilize the tibia.
  Other Names: intramedullary rodding
Procedure: surgery — combined surgery for enrolled patients with CPT: sleeve resection of the pathological soft tissues, retrograde intramedullary rodding, packaged lilac bone autograft,and llizarov external fixation device installation.
  Other Names: combined surgery

SUMMARY:
The study aims to evaluate the clinical result of Combined Surgery in Management of Congenital Pseudarthrosis.

DETAILED DESCRIPTION:
The study aims to evaluate the clinical result of Combined Surgery in Management of Congenital Pseudarthrosis. The combined surgery includes sleeve resection of the pathological soft tissues, retrograde intramedullary rodding, packaged lilac bone autograft,and appliance of llizarov external fixation device. Bone uion rate,average time of healing, Healing index, ankle valgus, limb length discrepancy, tibia axis alignment are recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria consists of patients with congenital pseudarthrosis of Tibia

Exclusion Criteria:

* Patients are complicated with mental, neurological disorders (such as hypoxic-ischemic encephalopathy, epilepsy and dementia) or significant barriers to growth.
* Patients with pseudarthrosis of tibia caused by trauma, tumor,infection, etc
* Children are complicated with dysfunction of liver and kidney , blood disorders, immune deficiency disease and ECG abnormalities.
* Parents refused further treatment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
whether the tibial has obtained union. | 6 months post-operation
  Ohnishi criterion: Degree of union was evaluated by the findings on radiographs and classified into three grades( Ohnishi criterion): union, delayed union, and nonunion. Radiographic union was defined as possessing continuity of bone density between the fragments without obvious radiolucent zone between them and possessing cortex-bridging fragments with sufficient thickness and radiodensity on both anteroposterior and lateral radiographs. Delayed union was defined as a process of healing that was slow but was progressing. Nonunion was defined by the healing process that had completely ceased.

SECONDARY OUTCOMES:
clinical outcome measurement(Johnston clinical evaluation criterion) | 3,6,9,12,18,24 months post-operation
  Johnston clinical evaluation criterion of Congenital Pseudarthrosis of Tibia (CPT): The outcome was classified as grade
  1 when there was unequivocal union with full weight-bearing function and maintenance of alignment requiring no additional surgical treatment; grade 2 when there was equivocal union with useful function, with the limb protected by a brace, and/or valgus or sagittal bowing for which additional surgery was required or anticipated; and grade 3 when there was persistent nonunion or refracture, requiring full-time external support for pain and/or instability.
Refracture of tibia | 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  The continuity of tibia cortex was disappeared in X ray.

OTHER OUTCOMES:
Residual Deformity-proximal tibia angulation(range,0°-90°) | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  measurement of the angulation of proximal tibia in anterior and posterior (AP )and lateral X ray
Residual Deformity-Limb length discrepancy | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  measurement of the length difference of both tibia in AP and lateral X ray
Residual Deformity-ankle valgus angulation(range,0°-90°) | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  measurement of the angulation between the distal tibia and ankle joint.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Yao, Principal Investigator — Hunan Children's Hospital
Locations (1):
- Hunan Children's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohnishi I, Sato W, Matsuyama J, Yajima H, Haga N, Kamegaya M, Minami A, Sato M, Yoshino S, Oki T, Nakamura K. Treatment of congenital pseudarthrosis of the tibia: a multicenter study in Japan. J Pediatr Orthop. 2005 Mar-Apr;25(2):219-24. doi: 10.1097/01.bpo.0000151054.54732.0b. PMID 15718906
- [Background] Romanus B, Bollini G, Dungl P, Fixsen J, Grill F, Hefti F, Ippolito E, Tudisco C, Wientroub S. Free vascular fibular transfer in congenital pseudoarthrosis of the tibia: results of the EPOS multicenter study. European Paediatric Orthopaedic Society (EPOS). J Pediatr Orthop B. 2000 Apr;9(2):90-3. doi: 10.1097/01202412-200004000-00003. PMID 10868357
- [Background] Johnston CE 2nd. Congenital pseudarthrosis of the tibia: results of technical variations in the charnley-williams procedure. J Bone Joint Surg Am. 2002 Oct;84(10):1799-810. PMID 12377911
- [Background] Malhotra D, Puri R, Owen R. Valgus deformity of the ankle in children with spina bifida aperta. J Bone Joint Surg Br. 1984 May;66(3):381-5. doi: 10.1302/0301-620X.66B3.6373777.
- [Background] Mathieu L, Vialle R, Thevenin-Lemoine C, Mary P, Damsin JP. Association of Ilizarov's technique and intramedullary rodding in the treatment of congenital pseudarthrosis of the tibia. J Child Orthop. 2008 Dec;2(6):449-55. doi: 10.1007/s11832-008-0139-4. Epub 2008 Oct 28. PMID 19308541
- [Derived] Zhu GH, Mei HB, He RG, Liu YX, Liu K, Tang J, Wu JY. Combination of intramedullary rod, wrapping bone grafting and Ilizarov's fixator for the treatment of Crawford type IV congenital pseudarthrosis of the tibia: mid-term follow up of 56 cases. BMC Musculoskelet Disord. 2016 Oct 22;17(1):443. doi: 10.1186/s12891-016-1295-1. PMID 27770774